CLINICAL TRIAL: NCT04010292
Title: Enhancing Patient Recall in Urogynecologic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, charbel salamon, PI/Medical Director of Urogynecology, Atlantic Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1448021-1
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Prolapse; Incontinence
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient education card (Experimental)
  Interventions: Behavioral: Patient education card
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Patient education card — Patient who are randomized to receive a patient card at the end of the counseling visit will be able to take an index-card sized card with them which will highlight their anticipated surgery.
  Arms: Patient education card

SUMMARY:
Patient counseling is an essential part of any new treatment implementation. This process becomes even more important when it involves surgical counseling. This is when the patient and the surgeon discuss the possible surgical options and ideally establish a plan for the appropriate surgical intervention. Unfortunately, multiple studies have shown that patients tend to have poor recall of the key elements discussed during the consultation (1-3). In the investigators' experience, the concern lies specifically in the level of recall that patients have regarding their planned surgical procedure, as most patients cannot correctly state the planned intervention despite extensive counseling and explanation. Lack of knowledge about the type of surgery can have serious implications for the patient in the future. For example, knowing facts like the presence or absence of the cervix and whether future pap smears are needed or the presence of an implant, such as a mesh are necessary for the patient's well-being and proper medical care down the line, especially when the patient has multiple medical providers. In addition, previous research has demonstrated that low-quality counseling and the feeling of being "unprepared for surgery" directly correlate with patient dissatisfaction (4). This is especially relevant in the field of female pelvic reconstructive surgery, where the success of surgical interventions relies heavily upon subjective patient-reported outcomes (5).

There have been many studies to augment the counseling process using supplemental materials. These have included use of multiple visual charts, anatomical models, and passive and interactive audiovisual aids (6). Some improvement in the outcomes has been observed in various fields of medicine with the dissemination of supplemental patient resources (7-10). However, in urogynecology, the effectiveness of surgical counseling sessions has not been achieved despite the different additional methods for patient education (6, 11). Reasons that urogynecologic supplemental materials have not seen the same level of success as those in other fields of medicine include the complexity of the surgeries and the language used in many of these educational aids (12). The investigators aim to address the problem of poor patient recall of their procedure by providing them with an easy-to-read patient card detailing the anticipated surgery at the time of their consult.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking females, ages >18 and <90 years, present for surgical planning for reconstructive urogynecologic procedures

Exclusion Criteria:

* Dementia, blindness, non-English speakers

Ages: 19 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient recall of the anticipated surgery during the preoperative visit | Patients will receive questionnaires within 30 days prior to their scheduled surgery.
  All patient present for a preoperative visit, which occurs within 30 days of the scheduled surgery. At this time, all patients will receive a questionnaire testing their knowledge about their upcoming surgery. We will compare the answers from patients who received the education card and those who did not at the time of their surgical counseling visit.
  The name of the questionnaire is "The 7-Question Knowledge Questionnaire," which was developed by the Urogynecology Department at Atlantic Health System. The scale consists of 7 questions and will have score ranges between from 0 to 7.

SECONDARY OUTCOMES:
Patient recall of the surgery during the postoperative visit | Patients will receive questionnaires within 30 days of their surgery.
  All patients will receive questionnaires, testing their knowledge of the performed surgery, during their postoperative follow-up visit.
  The questionnaire will include "The 7-Question Knowledge Questionnaire," which was developed by the Urogynecology Department at Atlantic Health System. The scale consists of 7 questions and will have score ranges between from 0 to 7.
Patient satisfaction | Patients will receive questionnaires within 30 days of their surgery.
  A validated questionnaire, called the "Leiden Perioperative care Patient Satisfaction questionnaire" will be given at the postoperative visit to determine patient satisfaction. A part of this questionnaire will be used, which consists of 4 questions. The total score will range between 0 and 4.

CONTACTS AND LOCATIONS:
Overall Officials: Charbel Salamon, MD, MS, Principal Investigator — Atlantic Health System
Locations (1):
- Atlantic Urogynecology Associates, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chernyak S, Caraballo R, Chiu S, Salamon C. Improving Patient Recall of Planned Intervention After Surgical Counseling: The IRIS Randomized Controlled Trial. Female Pelvic Med Reconstr Surg. 2022 May 1;28(5):280-286. doi: 10.1097/SPV.0000000000001102. Epub 2021 Sep 15. PMID 34534196